CLINICAL TRIAL: NCT05323565
Title: A Comparative Study Between the Use of Dexmedetomidine Versus Dexamethasone as Adjuvant to Bupivacaine in Ultrasound-guided Transversus Abdominis Plane Block for Post-operative Pain Relief in Patients Undergoing Lower Open Abdominal Surgeries
Brief Title: Dexmedetomine vs Dexamethasone in TAB Block for Abdominal Surgries
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Yasser Sayed Sobhy, Anesthesia specialist, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU M D 184/2020
Record Dates: First submitted 2022-04-05; First posted 2022-04-12 (Actual); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A (n=15): (Dexamethasone group) (Active Comparator): Patients will receive 20 ml 0.25% bupivacaine plus 4 mg dexamethasone on each side TAB bock.
  Interventions: Drug: Dexmedetomidine
- Group B (n=15): (Dexmedetomidine group) (Active Comparator): Patients will receive 20 ml 0.25% bupivacaine plus 0.5 mcg/kg of dexmedetomidine on each side TAB block.
  Interventions: Drug: Dexmedetomidine
- Group C (n=15): (control group) (Sham Comparator): Patients will receive 20 ml 0.25% bupivacaine on each side TAB block.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — adjuvants to 0.25 bupivacaine in TAB block.
  Other Names: dexamethasone

SUMMARY:
Randomized controlled clinical Trial to compare the efficacy and duration of postoperative analgesia achieved after adding dexmedetomidine or dexamethasone to bupivacaine in TAP block for lower open abdominal surgeries.

DETAILED DESCRIPTION:
A Comparative study between the use of dexmedetomidine versus dexamethasone as adjuvant to bupivacaine in ultrasound-guided transversus abdominis plane block for post-operative pain relief in patients undergoing lower open abdominal surgeries

ELIGIBILITY:
Inclusion Criteria:

Adult patients, Age 20-60 years. Elective operation under general anesthesia. Physical Status: ASA I and II Patients. Body mass index 25-35 kg/m2.

Exclusion Criteria:

* Infection at site of injection.
* Patient refusal.
* Psychiatric or physical illness that lead to inability to cooperate, speak or read.
* Abdominal operations under spinal anesthesia.
* History or evidence of coagulopathy.
* Known allergies to drugs used .
* Preexisting neurological disorders.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-07-05 (Estimated)

PRIMARY OUTCOMES:
1st time for rescue analgesia | first 24 hours post-operatively
  Time to first analgesia requirment(starting from drug injection)

SECONDARY OUTCOMES:
Pain score- Visual Analogue Score (VAS) | First 24 hours post-operatively.
  It ranges from 0 indicating no pain till 10 indicating severe intolerable pain with variable degrees of ascending pain in between] was assessed at 0 min (AT PACU), 2hr,6 hr, 12 hr, 18 hr, and 24 hr postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Yasser Sayed, Master, Principal Investigator — Ain Shams University, Faculty of medecine
Locations (1):
- Ain Shams University, Faculty of medicine, Cairo, Egypt